CLINICAL TRIAL: NCT01109238
Title: Trial Testing the Feasibility of Using Molecular-Guided Therapy in Patients With Refractory or Recurrent Neuroblastoma
Brief Title: A Trial Using Molecular-Guided Therapy in Patients With Refractory or Recurrent Neuroblastoma
Status: Completed | Type: Observational
Sponsor: Giselle Sholler (Other)
Collaborators: Van Andel Research Institute (Other)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Study Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Other Study IDs: NMTRC 001P
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Refractory Neuroblastoma; Relapsed Neuroblastoma
Keywords: Refractory Neuroblastoma; Relapsed Neuroblastoma
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Process Feasibility

SUMMARY:
The investigators are studying new ways to make treatment decisions for these types of cancer. Technologies at the Van Andel Research Institute (VARI) are available to determine a tumor's molecular makeup (gene expression profile). This technology (called "Xenobase") is being used to discover new ways to understand cancers and potentially predict the best treatments for patients with cancer. The researchers at VARI have filed a patent on the Xenobase and the specific network analysis method that the investigators will be using as part of this study.

A specimen obtained from the tumor during a recent surgical, biopsy, or bone marrow procedure will be sent to the Van Andel Research Institute. Researchers will attempt to identify the molecular makeup within the specimen, as well as in blood and urine samples in patients with aggressive and/or refractory cancer. This additional testing is different than the routine tests currently performed at the hospital for the evaluation of cancer.

The goals of this part of the study are: To determine if the investigators tumor board committee (at minimum a panel of 3 oncologists and 1 pharmacist) can use patient specific cancer cells to make real-time treatment decision using patient specific genetic information, and predicted therapies generated in the Xenobase report.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven neuroblastoma and confirmation of refractory or recurrent disease with histologic confirmation at diagnosis or at the time of recurrence/progression
* Patients must be age >12 months and diagnosed before the age of 21
* Life expectancy must be more than 3 months
* If measurable disease, this must be demonstrated by residual abnormal tissue at a primary or metastatic site measuring more than 1 cm in any dimension by standardized imaging (CT or MRI). For patients with only skeletal sites of disease, there must be at least one persisting focus with increased activity on a pre-treatment meta-iodobenzylguanidine (MIBG) scan.
* Current disease state must be one for which there is currently no known curative therapy
* Lansky Play Score must be more than 30
* Patients without bone marrow metastases must have an ANC > 750/μl and platelet count >50,000/μl
* Adequate liver function must be demonstrated, defined as:

  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age AND
  * SGPT (ALT) < 10 x upper limit of normal (ULN) for age
* No other significant organ toxicity defined as >Grade 2 by National Cancer Institute Common Toxicity Criteria for Adverse Events version 3 (NCI-CTCAE V3.0 (http://ctep.cancer.gov/forms/CTCAEv3.pdf))
* A negative serum pregnancy test is required for female participants of child bearing potential (≥13 years of age or after onset of menses)
* Both male and female post-pubertal study subjects need to agree to use one of the more effective birth control methods during treatment and for six months after treatment is stopped. These methods include total abstinence (no sex), oral contraceptives ("the pill"), an intrauterine device (IUD), levonorgestrol implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots). If one of these can not be used, contraceptive foam with a condom is recommended.
* Informed Consent: All patients and/or legal guardians must sign informed written consent. Assent, when appropriate, will be obtained according to institutional guidelines. Voluntary consent for optional biology studies will be included.

Exclusion Criteria:

* Patients who have received any chemotherapy within the last 21 days.
* Patients receiving anti-tumor therapy for their disease or any investigational drug concurrently
* Patients with serious infection or a life-threatening illness (unrelated to tumor) that is > Grade 2 (NCI CTCAE V3.0), or active, serious infections requiring parenteral antibiotic therapy within 2 weeks prior to screening
* Patients with any other medical condition, including malabsorption syndromes, mental illness or substance abuse, deemed by the Investigator to be likely to interfere with the interpretation of the results or which would interfere with a patient's ability to sign or the legal guardian's ability to sign the informed consent, and patient's ability to cooperate and participate in the study

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Relapsed and refractory Neuroblastoma
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of using protocol process to make real time treatment decisions | 4 months
  To pilot 5 patients to evaluate the feasibility of using predictive modeling based on genome-wide mRNA expression profiles of bone marrow derived neuroblastoma cells or tumor biopsies to make real-time treatment decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Sholler, MD, Study Chair — Beat Childhood Cancer at Atrium Health
Locations (1):
- UVM/FAHC, Burlington, Vermont, United States

REFERENCES:
- See also: Related Info — http://www.beatcc.org